CLINICAL TRIAL: NCT02287272
Title: Open-label, Randomized, Single Dose, 2-sequence, 2-period Cross-over Study to Investigate the Effect of Inhibition of the Organic Cation Transport in the Kidneys by Cimetidine on the Pharmacokinetics of the CHF5993 in Healthy Volunteers
Brief Title: Drug-drug Interaction Study of CHF5993 With Cimetidine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCD-05993AA1-12; 2013-005491-18 (EudraCT Number)
Record Dates: First submitted 2014-05-20; First posted 2014-11-10 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: COPD
Keywords: COPD- cimetidine- drug-drug interaction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Cimetidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment period R (Active Comparator): single inhaled dose of CHF 5993 pMDI (BDP/FF/GB fixed dose combination)
  Interventions: Drug: CHF 5993 pMDI
- Treatment period T (Active Comparator): Cimetidine plus CHF5993 pMDI: repeated doses of oral cimetidine for 6 days plus a single inhaled dose of CHF 5993 pMDI (BDP/FF/GB fixed dose combination)
  Interventions: Drug: Cimetidine plus CHF5993 pMDI

INTERVENTIONS:
Drug: CHF 5993 pMDI — 4 inhalations of CHF 5993 pMDI (BDP/FF/GB 100/6/25 micrograms per actuation) giving a total dose of 400, 24, 100 micrograms of BDP, FF, GB
  Arms: Treatment period R
Drug: Cimetidine plus CHF5993 pMDI — Cimetidine 800 milligrams twice daily for 6 days. On the fourth day, in addition, 4 inhalations of CHF5993 pMDI (BDP/FF/GB total dose 400/24/100 micrograms)
  Arms: Treatment period T

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic interaction when CHF5993 (pressurized metered-dose inhaler (pMDI) is administered with Cimetidine (probe inhibitor of the organic cation transport in the kidneys), by comparing the systemic exposure (AUC0-t) of Glycopyrronium Bromide (GB), after a single dose of the fixed combination CHF 5993 pMDI administered alone or at steady-state of Cimetidine

DETAILED DESCRIPTION:
the safety and tolerability of study treatments based on evaluation of vital signs, electrocardiograms and clinical laboratory assessments will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent obtained prior to any study-related procedure;
2. Male and female healthy volunteers aged 18-45 years inclusive;
3. Male subjects with female partner of childbearing potential: they or their partner must be willing to use (at least) one or more reliable methods of contraception (see exclusion criterion n.1 for details*) from the time of dose administration and until the end of the study. Male subjects must not donate sperm for 90 days after the last dose of study drug. Male subjects with partners of non-childbearing potential are not required to use contraception;
4. Able to understand the study procedures, the risks involved and ability to be trained to correctly use the devices;
5. Body Mass Index (BMI) between 18.0 and 30.0 kg/m2 inclusive;
6. A serum creatinine within the normal range (0,7-1,2 mg/dL) and an eGFR >80 mL/min/1.73 m2;
7. Non- or ex-smokers who smoked < 5 pack years (pack-years = the number of cigarette packs per day times the number of years) and stopped smoking > 1 year;
8. Good physical and mental status, determined on the basis of the medical history and a general clinical examination;

Exclusion Criteria:

1. Female subjects: pregnant or lactating women and all women physiologically capable of becoming pregnant (i.e. women of childbearing potential) UNLESS they meet the following definition of post-menopausal: 12 months of natural (spontaneous) documented amenorrhea or are willing to use one or more of the following reliable *methods of contraception:

   1. surgical sterilization (e.g. bilateral tubal ligation, hysterectomy for females; vasectomy for males)
   2. hormonal contraception (implantable, patch, oral), intrauterine device (IUD) or intrauterine system (IUS)
   3. barrier methods (male or female condom, diaphragm, sponge, cervical cap).
2. Blood donation (equal or more than 450 ml) or blood loss less than 8 weeks before inhalation of the study medication;
3. Positive HIV1 or HIV2 serology;
4. Positive results from the Hepatitis serology which indicates acute or chronic Hepatitis B or Hepatitis C;
5. History of substance abuse or drug abuse within 12 months prior to screening visit or with a positive urine drug screen at screening;
6. An abnormal triplicate 12-lead ECG (QRS> 120 msec, PR> 220 msec, HR < 40 bpm, HR > 110 bpm) at screening or at randomization;
7. Subjects whose electrocardiogram (12-lead ECG) shows QTcF >450 ms for males and >470 for females at screening or at randomization;
8. Subjects whose DBP is higher than 90 mmHg or SBP is higher than 140 mmHg at screening or at randomization;
9. Subjects who received any investigational new drug, or participated in clinical study within the last 8 weeks before screening;
10. History of hypersensitivity to M3 Antagonists, β2-agonist, corticosteroids or any of the excipients contained in any of the formulations used in the trial;
11. Treatment within the previous 3 months before the screening visit until the end of the study procedures in the last treatment period with any drug known to have a well-defined potential for hepatotoxicity (e.g. isoniazide, nimesulide, ketoconazole);
12. Subjects who refuse to abstain from alcohol or xanthine containing foods or beverages or grapefruit containing foods or beverages from 48 hour prior to each intake of study medication until the end of confinement at the clinical centre;
13. Heavy caffeine drinker (> 5 cups or glasses of caffeinated beverages e.g., coffee, tea, cola per day);
14. Subjects who have a positive urine test for cotinine at screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUC0-t) of Glycopyrronium Bromide | pre-dose, 5, 10,15,30min, 1,2,4,6,8,12hr post-dose

SECONDARY OUTCOMES:
Other pharmacokinetic parameters for Glycopyrronium Bromide | pre-dose-72hr post-dose
  Area under the plasma concentration-time curve from 0 to 72 hours (AUC0-72) and 0 hours to infinity (AUC0-inf); maximum concentration (Cmax), time to maximum concentration (tmax), and apparent systemic clearance (CL/F) of Glycopyrronium Bromide
Other pharmacokinetic parameters for Formoterol | pre-dose-24hr post dose
  Area under the plasma concentration-time curve from 0 to the last quantifiable concentration (AUC0-t), 0 to 24 hours (AUC0-24), 0 to 72 hours (AUC0-72) and 0 hours to infinity (AUC0-inf); maximum concentration (Cmax), time to maximum concentration (tmax), and apparent systemic clearance (CL/F) of Formoterol
Other pharmacokinetic parameters for B17MP | pre-dose- 72hr post-dose
  Area under the plasma concentration-time curve from 0 to the last quantifiable concentration (AUC0-t), 0 to 24 hours (AUC0-24), 0 to 72 hours (AUC0-72) and 0 hours to infinity (AUC0-inf); maximum concentration (Cmax), time to maximum concentration (tmax), and apparent systemic clearance (CL/F) of B17MP

CONTACTS AND LOCATIONS:
Overall Officials: Wouter Haazen, MD, Principal Investigator — Life Science Services SGS Belgium NV
Locations (1):
- Life Science Services SGS Belgium NV, Antwerp, Belgium

REFERENCES:
- [Result] Mariotti F, Ciurlia G, Spaccapelo L, Muraro A, Acerbi D. A Two-Period Open-Label, Single-Dose Crossover Study in Healthy Volunteers to Evaluate the Drug-Drug Interaction Between Cimetidine and Inhaled Extrafine CHF 5993. Eur J Drug Metab Pharmacokinet. 2017 Apr;42(2):269-279. doi: 10.1007/s13318-016-0345-2. PMID 27209586
- See also: CSR Synopsis available in the Chiesi Clinical Study Register — https://www.chiesi.com/clinic/CSR_Synopsis_CCD-05993AA1-12.pdf